CLINICAL TRIAL: NCT02388451
Title: The Benefits of the Use of the Feuerstein Cognitive Training Method on Cognitive Function in Community-dwelling Older Patients With Mild Cognitive Impairment: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 001
Record Dates: First submitted 2015-02-26; First posted 2015-03-17 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Feuerstein Program (Experimental): 15 subjects conforming to inclusion and exclusion criteria with a known clinical diagnosis of MCI and who provide informed consent will undergo cognitive and functional assessment to confirm the diagnosis of MCI. Baseline assessment using the Mindstreams Mild Cognitive Impairment Computerized Assessment Battery will be performed. Subjects will then participate 30 twice weekly meetings of 90 minutes duration each (for a total of 15 weeks). Mindstreams testing will be repeated after 15 sessions and at completion of the study.
  Interventions: Device: Feuerstein Program

INTERVENTIONS:
Device: Feuerstein Program — The IE activity is administered by instructors in groups of 10 to 15 participants. The intervention comprises 30 twice weekly meetings of 90 minutes duration per group.

SUMMARY:
15 subjects conforming to inclusion and exclusion criteria with a known clinical diagnosis of MCI and who provide informed consent will undergo cognitive and functional assessment to confirm the diagnosis of MCI. Baseline assessment using the Mindstreams Mild Cognitive Impairment Computerized Assessment Battery will be performed. Subjects will then participate 30 twice weekly meetings of 90 minutes duration each (for a total of 15 weeks). Mindstreams testing will be repeated after 15 sessions and at completion of the study.

DETAILED DESCRIPTION:
The rise in life expectancy in recent decades has resulted in a dramatic increase in the population of older people. This has been associated with a rise in the prevalence of age-associated conditions, particularly cognitive impairment and dementia. The prevalence of dementia in those older than 65 doubles every five years, and reaches a rate of more than 40% at age 85 years. Data from the World Health Organization predict 43 million dementia sufferers globally in the year 2020.

Mild Cognitive Impairment (MCI) is a syndrome comprising cognitive symptoms and impairment beyond population norms based on age and education, without functional loss. MCI represents a risk factor for dementia at a rate of conversion of approximately 12% annually. Thus patients with MCI characterize an important group for possible interventions in preventing further cognitive decline, particularly physical exercise and cognitive training.

The Feuerstein Program The Feuerstein Instrumental Enrichment (IE) program has been well-established as an effective intervention in other age groups and clinical situations. The method's creator, Professor Reuven Feuerstein, postulated that the thinking process is divided into three major phases - Input, Elaboration and Output - and that in each phase, different mental functions are at work. The quality of thinking depends upon the way the different functions are activated in each of the phases. The IE tools enable the correction or activation of cognitive deficiencies through use of targeted and focused mediation, which conserves and reinforces cognitive ability.

Recently, the Feuerstein Instrumental Enrichment Program for the Elderly was developed particularly for older people with cognitive decline.

Instrumental Enrichment can benefit all senior citizens, but is particularly recommended for those who do not constantly face intellectual challenges.

The process of learning IE is administered in group settings by instructors who have been trained to specifically mediate to the geriatric population. Work in groups constitutes a challenging, interesting and gratifying activity. It also appears that beyond contributing to the conservation and improvement of cognition, participating in the program may also have the effect of increasing feelings of competence, independence and improved emotional state.

15 subjects conforming to inclusion and exclusion criteria with a known clinical diagnosis of MCI and who provide informed consent will undergo cognitive and functional assessment to confirm the diagnosis of MCI. Baseline assessment using the Mindstreams Mild Cognitive Impairment Computerized Assessment Battery will be performed. Subjects will then participate 30 twice weekly meetings of 90 minutes duration each (for a total of 15 weeks). Mindstreams testing will be repeated after 15 sessions and at completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years and older
2. Able to read and speak Hebrew
3. Provide informed consent for participation in the study
4. Clinical diagnosis of MCI based on Consensus Criteria
5. A score of lower than 95 on the Memory Index of the Mindstreams Mild Cognitive Impairment Computerized Assessment Battery

Exclusion Criteria:

1. A medical condition (such as advanced heart failure, unstable ischemic heart disease, a lung condition with dyspnea on mild effort, intractable pain) or functional impairment (especially limiting mobility without the home) that does not allow the subject to participate in the training activities for the full duration of the study
2. A diagnosis of depression, bipolar disorder or schizophrenia
3. A cognitive diagnosis other than MCI, such as delirium, dementia or mental retardation
4. Visual impairment not corrected by the use of spectacles
5. Hearing impairment not corrected by hearing aids

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Mindstreams Mild Cognitive Impairment Computerized Assessment Battery | Change from Baseline Cognitive Function at 15 weeks
  The Mindstreams Mild Cognitive Impairment Computerized Assessment Battery developed by Neurotrax Corp. provides index scores in multiple cognitive domains, as well as a Global cognitive score

CONTACTS AND LOCATIONS:
Locations (1):
- Yan Press, Beersheba, Israel